CLINICAL TRIAL: NCT00918294
Title: QuickOptTM Study - Using the QuickOptTM Method for Timing Cycle Optimization
Acronym: QuickOpt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QuickOpt Study Asia
Record Dates: First submitted 2009-02-04; First posted 2009-06-11 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Heart Failure
Keywords: CRT; heart failure; optimization; Timing cycle optimization methods
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- QuickOpt (Experimental): QuickOpt is an optimization algorithm to program the AV, PV and VV delays
  Interventions: Device: QuickOpt

INTERVENTIONS:
Device: QuickOpt — The QuickOpt algorithm will suggest values for programming AV, PV and VV delay.

SUMMARY:
QuickOptTM optimization method provides a quicker, simpler and reliable alternative to standard echocardiography methods for optimization of sensed AV, paced AV and V-V delays in patients with CRT-P devices

ELIGIBILITY:
Inclusion Criteria:

* Patient meets current CRT-P indications and be implanted with an SJM CRT-P device with V-V timing and a compatible lead system
* Patient is able to provide written informed consent for study participation

Exclusion Criteria:

* Patient has limited intrinsic atrial activity (≤ 40 bpm)
* Patient has persistent or permanent AF
* Patient has a 2o or 3o heart block
* Patient is unable to provide analyzable echocardiogram images
* Patient's life expectancy is <12 months
* Patient is <18 years old
* Patient is pregnant
* Patient is on IV inotropic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To compare the aortic velocity time integral value derived by the QuickOptTM optimization method with that derived by the standard echocardiography optimization methods | 1 day

SECONDARY OUTCOMES:
Time required for each optimization method considered in this study | 1 day
Effects of any spontaneous cardiac events during the QuickOpt optimization process and these events are not limited to premature ventricular complex (PVC), pacemaker-mediated tachycardia (PMT), atrial fibrillation (AF) and far-field R-wave oversensing | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Fu Wai Hospital, Beijing, China

REFERENCES:
- [Derived] Hua W, Wang DM, Cai L, Sun CF, Fu GS, Wang YT, Yan J, Luo ZL, Xu J, Wang ZY, Xu G, Shen FR, Xu W, Wang JF, Ren XJ, Jin W, Zhang N, Lau EO, Zhang S. A prospective study to evaluate the efficacy of an intracardiac electrogram-based atrioventricular and interventricular intervals optimization method in cardiac resynchronization therapy. Chin Med J (Engl). 2012 Feb;125(3):428-33. PMID 22490397